CLINICAL TRIAL: NCT03152630
Title: Research on the Early and Prognosis Diagnosis of Vascular Dementia
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201512101RINA
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Dementia
Keywords: lncRNAs; Alzheimer's disease; vascular dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Around 10% of stroke survivors develop dementia within 3 months after stroke and over 20% more stroke patients have dementia in the subsequent 3 years. Previous studies documented a close relationship between stroke and Alzheimer's disease (AD). There are, however, no reliable biomarkers to detect cognitive dysfunction and dementia among stroke patients or to predict the risks of vascular dementia (VD) and AD among patients with stroke. There is a clear need to identify novel mediators of cognitive dysfunction in stroke patients to provide insights into the pathogenesis, to tailor clinical care based on risks, and to develop new therapeutic strategies.

While the expression of messenger RNAs (mRNAs) and microRNAs (miRNAs) account for only ~1% of all transcribed species, up to 90% of the mammalian genome is transcribed as long non-coding RNAs (lncRNAs), a heterogeneous group of non-coding transcripts longer than 200 nucleotides. LncRNAs have been shown to be functional and involved in specific physiological and pathological processes through epigenetic, transcriptional and post-transcriptional mechanisms. While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to cognitive dysfunction and dementia in stroke patients.

In this proposal, we seek to apply next-generation sequencing technology to investigate circulating lncRNA expression, as well as exosomal RNAs in the subjects with and without cognitive dysfunction or dementia. In addition, we will apply the near-infrared spectroscopy (NIRS) to evaluate cerebral blood flow, metabolism and oxygenation in these subjects. We will test the hypothesis that circulating lncRNA/exosomal RNA signature and NIRS imagaing can reflect the cognitive states in stroke patients. The accuracy, sensitivity and specificity of the lncRNA-exosomal RNA-NIRS-based cognitive dysfunction scoring system will then be tested in an independent, large validation cohort. Next, we propose to test the hypothesis that circulating lncRNAs/exosomal RNA and NIRS imaging can be novel prognostic biomarkers to predict cognitive dysfunction and dementia in stroke patients. These studies will also establish a set of novel, lncRNA-based diagnostic and prognostic biomarker in stroke patients to improve clinical preventive and therapeutic care.

DETAILED DESCRIPTION:
Around 10% of stroke survivors develop dementia within 3 months after stroke and over 20% more stroke patients have dementia in the subsequent 3 years. Previous studies documented a close relationship between stroke and Alzheimer's disease (AD). There are, however, no reliable biomarkers to detect cognitive dysfunction and dementia among stroke patients or to predict the risks of vascular dementia (VD) and AD among patients with stroke. There is a clear need to identify novel mediators of cognitive dysfunction in stroke patients to provide insights into the pathogenesis, to tailor clinical care based on risks, and to develop new therapeutic strategies.

It has become increasingly clear that the transcription of the eukaryotic genome is far more pervasive and complex than previously appreciated. While the expression of messenger RNAs (mRNAs) and microRNAs (miRNAs) account for only ~1% of all transcribed species, up to 90% of the mammalian genome is transcribed as long non-coding RNAs (lncRNAs), a heterogeneous group of non-coding transcripts longer than 200 nucleotides. LncRNAs have been shown to be functional and involved in specific physiological and pathological processes through epigenetic, transcriptional and post-transcriptional mechanisms. While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to cognitive dysfunction and dementia in stroke patients. Exosomes are small vesicles of endocytic origin that are released into the extracellular environment and may participate in signal transduction between cells. Exosomes from central nervous system can penetrate blood brain barrier and can be collected from serum. Recently, exosomes had been shown containing several kinds of important protein and RNA and played roles in post diseased cell survival and death. Our previous studies focus on the specific inflammatory responses in neurons receiving ischemic injury. We have used blood samples in acute stroke patients to verify the relationship between specific signaling proteins in inflammatory pathways and post stroke functional outcome. Besides, our ongoing project also found that exosomes released from neurons with oxygen glucose deprivation may be related to the post stroke inflammation.

NIR spectroscopy is a revolutionary new device allowing the measurement of oxygenated and de-oxygenated hemoglobin concentrations in tissue. The device works by emitting Near Infrared (NIR) light into tissue at known diffusion path from a detector. Once the absorption and scattering are determined, the assumption that hemoglobin is the only significant absorber is applied and the oxygenated and de-oxygenated hemoglobin concentrations are calculated. The applications of the NIR spectroscopy include but are not limited to Peripheral Vascular Disease, Cardiothoracic & Vascular Surgery, and Neurosurgery. We have also developed a prototype of near-infrared spectroscopy. The preliminary findings and possible clinical value of this technology has been proven.

In this proposal, we seek to apply next-generation sequencing technology to investigate circulating lncRNA expression, as well as exosomal RNAs in the subjects with and without cognitive dysfunction or dementia. In addition, we will apply the near-infrared spectroscopy (NIRS) to evaluate cerebral blood flow, metabolism and oxygenation in these subjects. We will test the hypothesis that circulating lncRNA/exosomal RNA signature and NIRS imagaing can reflect the cognitive states in stroke patients. The accuracy, sensitivity and specificity of the lncRNA-exosomal RNA-NIRS-based cognitive dysfunction scoring system will then be tested in an independent, large validation cohort. Next, we propose to test the hypothesis that circulating lncRNAs/exosomal RNA and NIRS imaging can be novel prognostic biomarkers to predict cognitive dysfunction and dementia in stroke patients. These studies will also establish a set of novel, lncRNA-based diagnostic and prognostic biomarker in stroke patients to improve clinical preventive and therapeutic care.

ELIGIBILITY:
Inclusion Criteria:

* age older than 20 years old
* willing to sign ICF
* report oneself disease
* have Taiwanese ID
* atherosclerotic vascular diseases, but with at least 1 CV risk factor [DM, dyslipidemia or under lipid lowering therapy, hypertension, smoking, old (M>45, F>55 years), family history of premature CAD, obesity

Exclusion Criteria:

* not willing to sign ICF

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: In this project, three hundred male or female patients with stable symptomatic atherosclerotic disease over 20 years of age will be enrolled from our previous registry program. Peripheral atherosclerosis with symptoms of ischemia and confirmed by ankle-brachial index, Doppler ultrasound, or angiography will also be included (group A). The other 600 patients will be enrolled with no evidence of atherosclerotic vascular diseases, but with at least 1 CV risk factor [DM, dyslipidemia (TC >200 mg/dL; LDL-C > 130 mg/dL ; TG > 200 mg/dL; male HDL-C < 40 mg/dL ; female HDL-C < 50 mg/dL) or under lipid lowering therapy, hypertension, smoking, old (M>45, F>55 years), family history of premature CAD (M<55, F<65 years), obesity (waist: M>90, F>80 cm)] (group B).
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-03-30 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | up to 5 years
  The composite cardiovascular (CV) outcome will be any CV events (coronary, cerebral, or peripheral vascular diseases)

SECONDARY OUTCOMES:
With at least 1 cardiovascular risk factor. | up to 5 years
  no evidence of atherosclerotic vascular diseases,with at least 1 cardiovascular risk factor.

CONTACTS AND LOCATIONS:
Overall Officials: Chau C Wu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes